CLINICAL TRIAL: NCT00092274
Title: An Open-label, International, Multicenter, Dose Escalating, Phase I/II Study of HuMax-CD20 in Patients With Relapsed or Refractory Follicular Lymphoma Grade I-II
Brief Title: Study of HuMax-CD20, a New Drug to Treat Early Stage Non-Hodgkin´s Follicular Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Acquired asset
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hx-CD20-001
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2005-01

CONDITIONS: Lymphoma, Follicular
Keywords: Follicular Lymphoma; Non Hodgkin´s Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — ofatumumab

INTERVENTIONS:
Drug: HuMax-CD20

SUMMARY:
The purpose of this trial is to determine the safety and efficacy of HuMax-CD20 as a treatment for Follicular Lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory follicular lymphoma grade I-II
* Tumor verified to be CD20 positive
* CT scan showing demarcated lesions

Exclusion Criteria:

* Previous treatment with rituximab resulting in less than partial response
* Previous radioimmunotherapy
* Previous stem cell transplantation
* Received the following treatments within 4 weeks prior to entering this study:

  1. Anti-cancer therapy
  2. Glucocorticosteroids unless less than 10 mg prednisolone/day
  3. Radiotherapy
* Received Mitomycin C or Nitrosoureas within 6 weeks prior to entering this trial
* HIV positivity
* Hepatitis B or hepatitis C
* Uncontrolled or chronic bacterial, fungal or viral infection
* Other cancer diseases, except certain skin cancers, cervix cancer and breast cancer
* Certain serious medical conditions, including kidney or liver disease, some psychiatric illnesses, and stomach, lung, heart, hormonal, nerve or blood diseases
* WHO performance status of 3 or 4
* If you are participating in another trial with a different new drug 4 weeks before you enter this trial
* Current participation in any other clinical study
* Pregnant or breast-feeding women
* Women of childbearing age who are unable or unwilling to use an IUD or hormonal birth control during the whole trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-09; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Struemper H, Sale M, Patel BR, Ostergaard M, Osterborg A, Wierda WG, Hagenbeek A, Coiffier B, Jewell RC. Population pharmacokinetics of ofatumumab in patients with chronic lymphocytic leukemia, follicular lymphoma, and rheumatoid arthritis. J Clin Pharmacol. 2014 Jul;54(7):818-27. doi: 10.1002/jcph.268. Epub 2014 Jan 28. PMID 24443277
- [Derived] Hagenbeek A, Gadeberg O, Johnson P, Pedersen LM, Walewski J, Hellmann A, Link BK, Robak T, Wojtukiewicz M, Pfreundschuh M, Kneba M, Engert A, Sonneveld P, Flensburg M, Petersen J, Losic N, Radford J. First clinical use of ofatumumab, a novel fully human anti-CD20 monoclonal antibody in relapsed or refractory follicular lymphoma: results of a phase 1/2 trial. Blood. 2008 Jun 15;111(12):5486-95. doi: 10.1182/blood-2007-10-117671. Epub 2008 Apr 4. PMID 18390837